CLINICAL TRIAL: NCT00308256
Title: Effects of Nurse-counselling in the Improvement of the type1 Diabetes Control in Adolescents: a Randomized Controlled Trial
Brief Title: Effects of Nurse-counselling in the Improvement of the type1 Diabetes Control in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2005.395
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
Keywords: Type1 diabetes;; nurse-counselling;; adolescent
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (2):
- Nurse counseling (Experimental): Phone calls performed by nurse 15 days after each monthly visit
  Interventions: Behavioral: nurse-counselling
- Control (No Intervention): Normal monthly follow-up without phone calls

INTERVENTIONS:
Behavioral: nurse-counselling — Phone calls performed by nurse 15 days after each monthly visit
  Arms: Nurse counseling

SUMMARY:
The incidence of type 1 diabetes is increasing in France. A recent cross sectional study has shown that in France, only 15% of children and 26% of adults had HbA1c<7%. Adolescents seem to need particularly a better metabolic control.

Working Hypothesis:

We hypothesized that a stricter control of glycaemia by nurse-counselling could probably improve metabolic control in adolescents with type 1 diabetes.

Objectives:

To show that nurse-counselling may improve levels of patient satisfaction.

Methodology:

The main criterion is the patient acceptance of diabetes measured by an analogical visual scale rated from 0 (I cope very well with my diabetes, I cope very badly with my diabetes) to 10 cm. The scale will be measured every quarter within 12 months follow-up. We wish to improve patient's appreciation by 10 mm, near to "I cope very well with my diabetes".

This is a randomised parallel group study with 36 subjects in each group. During the follow-up, the "routine follow-up" group will continue its routine care. The "complementary follow-up" group will be called by nurses every 15 days and consult monthly. HbA1c is the secondary criterion and will be measured every 3 months.

The total study duration is 18 months including 6 months for the recruitment and 12 months for the patients follow-up

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 13 to 18 years with a type1 diabetes diagnosed at least one year earlier,
* HbA1c rate > 8 %.

Exclusion Criteria:

* HbA1c < 8 %;
* patients participating in another study

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2006-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Patient's acceptance of the disease evaluated by an analogical visual scale rating | 12 months

SECONDARY OUTCOMES:
Glycaemic equilibrium by measuring the rate of glycosylated haemoglobin | 12 months
Number of diabetic acidosis having required hospitalization, | 12 months
Episodes number of severe hypoglycaemia having required an intervention of a third party or a hospitalization. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc NICOLINO, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Marc Nicolino, Lyon, France

REFERENCES:
- [Result] Kassai B, Rabilloud M, Bernoux D, Michal C, Riche B, Ginhoux T, Laudy V, Terral D, Didier-Wright C, Maire V, Dumont C, Cottancin G, Plasse M, Jeannoel GP, Khoury J, Bony C, Lievre M, Drai J, Nicolino M. Management of adolescents with very poorly controlled type 1 diabetes by nurses: a parallel group randomized controlled trial. Trials. 2015 Sep 8;16:399. doi: 10.1186/s13063-015-0923-7. PMID 26350209